CLINICAL TRIAL: NCT06709092
Title: Study on the Effect and Mechanism of Lupatadine Fumarate in the Treatment of Allergic Rhinitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng Lei (Other)
Responsible Party: Sponsor-Investigator, Cheng Lei, chief physician, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-674
Record Dates: First submitted 2024-01-21; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Allergic rhinitis (Experimental): For patients with AR, patients were given lupatadine fumarate (Luso®, Yangzijiang Pharmaceuticals) 1 tablet once daily at bedtime for 14 days.
  Interventions: Drug: lupatadine fumarate (Luso®, Yangzijiang Pharmaceuticals)

INTERVENTIONS:
Drug: lupatadine fumarate (Luso®, Yangzijiang Pharmaceuticals) — For patients with AR, patients were given lupatadine fumarate (Luso®, Yangzijiang Pharmaceuticals) 1 tablet once daily at bedtime for 14 days.

SUMMARY:
In China, the prevalence of allergic rhinitis reaches 17.6% and is increasing year by year, seriously affecting the quality of life of patients. Some patients still cannot be effectively treated. So it is urgent to study the pathogenesis of AR and find new therapeutic targets. Lupatadine fumarate has the dual effects of antihistamine and platelet-activating factor (PAF), and it is the only potent and highly effective allergy drug with both antihistamine and PAF antagonism currently on the marke. The exact mechanism of Lupatadine fumarate in relieving nasal congestion in patients with AR is unknown. Tight junction proteins (TJs) play an important role in maintaining endothelial barrier function, and TJ disruption disrupts barrier function and promotes inflammation. 15-LOX(15-lipoxygenase) disrupts tight junctions at the blood-brain barrier. It increases cerebral vascular permeability and contributes to cerebral edema. In a mouse model of atherosclerosis, 15(S)-HETE, the major metabolite of 15-LOX, enhances the phosphorylation of ZO-2 at the Thr-1/1 residue through MEK1-ERK770/772 activation, leading to the dissociation of ZO-1 from occludin and disrupting the endothelial TJ and its barrier function. So we want to study the effects and mechanisms of lupatadine fumarate in the treatment of allergic rhinitis (AR) and whether lupatadine fumarate is directly related to 15-LO1.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-65 years).
* Patients with allergic rhinitis were diagnosed based on clinical history and positive dust mite sensitization tests (skin prick test and/or specific IgE).

Exclusion Criteria:

* Received glucocorticoids, immunomodulatory, antihistamine drugs, and other medications that may affect the study results within the last 1 month.
* Nasal diseases such as upper respiratory tract infections, chronic sinusitis with or without nasal polyps, and nasal sinus tumors.
* History of nasal sinus surgery.
* With other immune and allergic diseases.
* Patients with a combination of severe cardiac, cerebrovascular or pulmonary - diseases, aspirin triad, primary ciliary dyskinesia, immune deficiency, and coagulation disorders.
* Pregnant women.
* Smokers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rhinoconjunctivitis Quality of Life Questionnaire | baseline and 14 days
  To measure the functional impairments that are most troublesome to adult patients as a result of their rhinoconjunctivitis. Patients were scored by questionnaire before and after treatment, and the change in score before and after treatment was the primary outcome measure. 7-point scale (0 = not impaired at all - 6 = severely impaired). Higher scores reflect lower quality of life.
Visual analogue scale | baseline and 14 days
  Results VAS are well validated for the measurement of AR symptoms and correlate well with the ARIA (allergic rhinitis and its impact on asthma) severity classification. Patients were scored by questionnaire before and after treatment, and the change in score before and after treatment was the primary outcome measure. Range: 0-10. Higher scores reflect more pain and severity.
The concentration of interleukin 4(IL-4), interleukin 5(IL-5), interleukin 13(IL-13) | baseline and 14 days
  It reflects Th2 immune response in patients with allergic rhinitis

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Al-Digheari A, Mahboub B, Tarraf H, Yucel T, Annesi-Maesano I, Doble A, Lahlou A, Tariq L, Aziz F, El Hasnaoui A. The clinical burden of allergic rhinitis in five Middle Eastern countries: results of the SNAPSHOT program. Allergy Asthma Clin Immunol. 2018 Nov 19;14:63. doi: 10.1186/s13223-018-0298-x. eCollection 2018. PMID 30473712
- [Background] Eifan AO, Durham SR. Pathogenesis of rhinitis. Clin Exp Allergy. 2016 Sep;46(9):1139-51. doi: 10.1111/cea.12780. PMID 27434218
- [Background] Cheng L, Chen J, Fu Q, He S, Li H, Liu Z, Tan G, Tao Z, Wang D, Wen W, Xu R, Xu Y, Yang Q, Zhang C, Zhang G, Zhang R, Zhang Y, Zhou B, Zhu D, Chen L, Cui X, Deng Y, Guo Z, Huang Z, Huang Z, Li H, Li J, Li W, Li Y, Xi L, Lou H, Lu M, Ouyang Y, Shi W, Tao X, Tian H, Wang C, Wang M, Wang N, Wang X, Xie H, Yu S, Zhao R, Zheng M, Zhou H, Zhu L, Zhang L. Chinese Society of Allergy Guidelines for Diagnosis and Treatment of Allergic Rhinitis. Allergy Asthma Immunol Res. 2018 Jul;10(4):300-353. doi: 10.4168/aair.2018.10.4.300. PMID 29949830
- [Background] Ren Q, Ren L, Ren C, Liu X, Dong C, Zhang X. Platelet endothelial cell adhesion molecule-1 (PECAM1) plays a critical role in the maintenance of human vascular endothelial barrier function. Cell Biochem Funct. 2015 Dec;33(8):560-5. doi: 10.1002/cbf.3155. Epub 2015 Nov 25. PMID 26607202
- [Background] Soon AS, Chua JW, Becker DL. Connexins in endothelial barrier function - novel therapeutic targets countering vascular hyperpermeability. Thromb Haemost. 2016 Oct 28;116(5):852-867. doi: 10.1160/TH16-03-0210. Epub 2016 Aug 4. PMID 27488046
- [Background] Cong X, Kong W. Endothelial tight junctions and their regulatory signaling pathways in vascular homeostasis and disease. Cell Signal. 2020 Feb;66:109485. doi: 10.1016/j.cellsig.2019.109485. Epub 2019 Nov 23. PMID 31770579